CLINICAL TRIAL: NCT01188499
Title: A Phase 1B/2A, Open-label, Non-randomized, Multi-arm Study of TL32711 in Combination With Chemotherapy in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Dose Escalation, Combination Chemotherapy Safety Study of Birinapant (TL32711), in Subjects With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TetraLogic Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TL32711-POC-0078-PTL
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — birinapant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Carboplatin/Paclitaxel + Birinapant (Experimental): Carboplatin (AUC 6/Paclitaxel (175 mg/m2/IV) once every 3 (q3) weeks + birinapant (TL32711) once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  Interventions: Drug: Birinapant
- Irinotecan + Birinapant (Experimental): Irinotecan (350 mg/m2/IV) once every 3 (q3) weeks + birinapant (TL32711) once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  Interventions: Drug: Birinapant
- Docetaxel + Birinapant (Experimental): Docetaxel (75 mg/m2/IV) once every 3 (q3) weeks + birinapant (TL32711) once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  Interventions: Drug: Birinapant
- Gemcitabine + Birinapant (Experimental): Gemcitabine (1000 mg/m2/IV) once weekly (7 days +/- 2 days) for 3 consecutive weeks followed by 1 week off + birinapant (TL32711) once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 2 week off for each cycle (4 weeks per cycle).
  Interventions: Drug: Birinapant
- Liposomal Doxorubicin + Birinapant (Experimental): Liposomal doxorubicin (40 mg/m2/IV) every 4 weeks + birinapant (TL32711) once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 2 weeks off for each cycle (4 weeks per cycle).
  Interventions: Drug: Birinapant

INTERVENTIONS:
Drug: Birinapant
  Other Names: TL32711

SUMMARY:
This is a dose escalation safety study of birinapant (TL32711) in combination with chemotherapy in subjects with advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety and maximum tolerated dose of birinapant (TL32711) as a 30 minute intravenous infusion once a week, for 2 consecutive weeks, when combined with standard regimens of chemotherapy in subjects with advanced or metastatic solid tumors. Additionally the study will assess anti-tumor activity, pharmacokinetics, and exploratory biomarkers as a measurement of pharmacodynamic effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed advanced or metastatic malignancy for which the proposed chemotherapy regimen is appropriate in the judgment of the Investigator.
* Prior therapy in dose-escalation and expansion cohorts:

  * Dose-escalation cohorts: Subjects may be naïve or may have received prior therapy with the specific chemotherapeutic agent(s) being recommended in the combination arm, provided the subject did not experience life-threatening toxicity attributed to the specific agent(s).
  * Expansion cohorts: Subjects have advanced colorectal cancer that had been previously determined to be KRAS mutant. Subjects naïve to irinotecan may be enrolled, and the KRAS mutation status may be wild type or mutant. Subjects previously treated with an irinotecan containing regimen may be enrolled only if they have been previously determined to be KRAS wild type. The irinotecan regimen must not have been associated with life threatening adverse events.
* Subjects evaluated for Arm 5 (liposomal doxorubicin) may not have received >300 mg/m2 cumulative dose of anthracycline.
* Life expectancy >3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* Adequate renal function
* Adequate hepatic function
* Adequate bone marrow function
* Women of childbearing potential must have a negative serum pregnancy test.
* Women of childbearing potential must agree to use 2 methods of adequate contraception (ie, hormonal and barrier method) prior to enrollment, during the study, and for a period of 30 days following the last dose of TL32711. Males who are sexually active must agree to use a condom during the study and for a period of 30 days following the last dose of TL32711, and if their partner is of childbearing potential, she must agree to use a secondary method of contraception (ie, hormonal, intrauterine device, barrier) during the study and for a period of 30 days following the last dose of TL32711.

Exclusion Criteria:

* Recent anti-cancer treatment defined as:

  * Standard or investigational anti-cancer therapy within 4 weeks prior to first dose of TL32711. Exception: continued hormonal interventions for prostate cancer.
  * Radiation therapy within 2 weeks prior to the first dose of TL32711.
  * Major surgery within 4 weeks prior to the first dose of TL32711. Subjects must be well recovered from acute effects of surgery prior to enrollment.
* Known or suspected diagnosis of human immunodeficiency virus or chronic active Hepatitis B or C.
* Symptomatic or uncontrolled brain metastases requiring current treatment.
* Impaired cardiac function or clinically significant cardiac disease
* QT interval corrected for heart rate (QTcB) >480 msec (including subjects on medication).
* Lack of recovery of prior adverse events to Grade ≤1 severity (NCI CTCAE v4) (except alopecia) due to therapy administered prior to the initiation of study drug dosing.
* Nursing or pregnant women.
* Known allergy to any of the formulation components of TL32711.
* Any concurrent disease and/or medical condition that in the opinion of the Investigator that would prevent the subject's participation, render the subject at excessive risk (including excessive risks due to the toxicity profile of the planned combination chemotherapeutic regimen), or limit the subject's compliance with the protocol's required evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-10; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John N Nemunaitis, MD, Principal Investigator — Mary Crowley Cancer Research Center; Ravi Amaravadi, MD, Principal Investigator — University of Pennsylvania, Abramson Cancer Center; Lainie P Martin, MD, Principal Investigator — Fox Chase Cancer Center; Alex Adjei, MD, PhD, Principal Investigator — Roswell Park Cancer Institute; Patricia LoRusso, DO, Principal Investigator — Barbara Ann Karmanos Cancer Center; Kyriakos P Papadopoulos, MD, Principal Investigator — South Texas Accelerated Research Therapeutics (START); Zdenka Segota, MD, Principal Investigator — Holy Cross Hospital
Locations (7):
- United States (7):
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Carboplatin/Paclitaxel + Birinapant: Carboplatin (AUC 6/Paclitaxel (175 mg/m2/IV) once every 3 (q3) weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by one week off repeated every 3 weeks as tolerated in combination with chemotherapy
- Arm 2: Irinotecan + Birinapant: Irinotecan (350 mg/m2/IV) once every 3 (q3) weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by one week off repeated every 3 weeks as tolerated in combination with chemotherapy
- Arm 3: Docetaxel + Birinapant: Docetaxel (75 mg/m2/IV) once every 3 (q3) weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by one week off repeated every 3 weeks as tolerated in combination with chemotherapy
- Arm 4: Gemcitabine + Birinapant: Gemcitabine (1000 mg/m2/IV) once weekly (7 days +/- 2 days) for 3 consecutive weeks followed by 1 week off + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 2 week off for each cycle (4 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by two weeks off repeated every 4 weeks as tolerated in combination with chemotherapy.
- Arm 5: Liposomal Doxorubicin + Birinapant: Liposomal doxorubicin (40 mg/m2/IV) every 4 weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 2 weeks off for each cycle (4 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by two weeks off repeated every 4 weeks as tolerated in combination with chemotherapy.
Period: Overall Study
Arm/Group | Arm 1: Carboplatin/Paclitaxel + Birinapant | Arm 2: Irinotecan + Birinapant | Arm 3: Docetaxel + Birinapant | Arm 4: Gemcitabine + Birinapant | Arm 5: Liposomal Doxorubicin + Birinapant
Started | 24 | 83 | 33 | 18 | 18
Completed | 24 | 83 | 33 | 18 | 18
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Carboplatin/Paclitaxel + Birinapant | Arm 2: Irinotecan + Birinapant | Arm 3: Docetaxel + Birinapant | Arm 4: Gemcitabine + Birinapant | Arm 5: Liposomal Doxorubicin + Birinapant | Total
Number analyzed (Participants) | 24 | 83 | 33 | 18 | 18 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8.77) | 59.6 (11.58) | 60.7 (11.16) | 56.7 (8.55) | 56.5 (10.44) | 59.7 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 39 | 15 | 11 | 13 | 91
  Male | 11 | 44 | 18 | 7 | 5 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 2 | 2 | 8
  Not Hispanic or Latino | 23 | 81 | 32 | 16 | 16 | 168
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 12 | 3 | 3 | 3 | 23
  White | 22 | 71 | 30 | 15 | 13 | 151
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 24 | 83 | 33 | 18 | 18 | 176

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events as a Measure of Safety and Tolerability
Description: Number of subjects with adverse events as a measure of safety and tolerability including changes in vital signs, electrocardiograms (ECGs), safety and laboratory parameters
Time Frame: 1 Cycle (3-4 weeks)
Measure: Number; unit: participants
Groups:
- Arm 1: Carboplatin/Paclitaxel + TL32711: Carboplatin (AUC 6/Paclitaxel (175 mg/m2/IV) once every 3 (q3) weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by one week off repeated every 3 weeks as tolerated in combination with chemotherapy
- Arm 2: Irinotecan + TL32711: Irinotecan (350 mg/m2/IV) once every 3 (q3) weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by one week off repeated every 3 weeks as tolerated in combination with chemotherapy
- Arm 3: Docetaxel + TL32711: Docetaxel (75 mg/m2/IV) once every 3 (q3) weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 1 week off for each cycle (3 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by one week off repeated every 3 weeks as tolerated in combination with chemotherapy
- Arm 4: Gemcitabine + TL32711: Gemcitabine (1000 mg/m2/IV) once weekly (7 days +/- 2 days) for 3 consecutive weeks followed by 1 week off + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 2 week off for each cycle (4 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by two weeks off repeated every 4 weeks as tolerated in combination with chemotherapy.
- Arm 5: Liposomal Doxorubicin: Liposomal doxorubicin (40 mg/m2/IV) every 4 weeks + TL32711 once weekly (7 days +/- 2 days) for 2 consecutive weeks followed by 2 weeks off for each cycle (4 weeks per cycle).
  TL32711: 30 minute intravenous (IV) infusion of TL32711 administered once weekly for two consecutive weeks followed by two weeks off repeated every 4 weeks as tolerated in combination with chemotherapy.
Arm/Group | Arm 1: Carboplatin/Paclitaxel + TL32711 | Arm 2: Irinotecan + TL32711 | Arm 3: Docetaxel + TL32711 | Arm 4: Gemcitabine + TL32711 | Arm 5: Liposomal Doxorubicin
Number analyzed (Participants) | 24 | 83 | 33 | 18 | 18
participants | 24 | 83 | 33 | 18 | 18
Statistical Analysis 1: Comparison: Arm 1: Carboplatin/Paclitaxel + TL32711 vs Arm 2: Irinotecan + TL32711 vs Arm 3: Docetaxel + TL32711 vs Arm 4: Gemcitabine + TL32711 vs Arm 5: Liposomal Doxorubicin; Test type: Superiority or Other; Percent = 100 — Primary objective of safety and tolerability measured by percent participants experiencing at least one adverse event. No formal statistics performed

2. Secondary Outcome: Evaluation of Anti-tumor Efficacy
Description: Tumor burden according to Response Evaluation Criteria in Solid Tumors (RECIST) and time to progression
Time Frame: Every 2 cycles
Population: Intent-to-treat (ITT)
Measure: Number; unit: participants
Arm/Group | Arm 1: Carboplatin/Paclitaxel + TL32711 | Arm 2: Irinotecan + TL32711 | Arm 3: Docetaxel + TL32711 | Arm 4: Gemcitabine + TL32711 | Arm 5: Liposomal Doxorubicin
Number analyzed (Participants) | 24 | 83 | 33 | 18 | 18
participants | 5 | 8 | 3 | 2 | 0
Statistical Analysis 1: Comparison: Arm 1: Carboplatin/Paclitaxel + TL32711 vs Arm 2: Irinotecan + TL32711 vs Arm 3: Docetaxel + TL32711 vs Arm 4: Gemcitabine + TL32711 vs Arm 5: Liposomal Doxorubicin; Test type: Superiority or Other; Percent = 10 — Percent patients overall across all five arms demonstrating complete or partial response by RECIST. No formal statistics performed

3. Secondary Outcome: Evaluation of Pharmacokinetics and Translational Biomarkers
Description: Measurement of TL32711 pharmacokinetics: Maximum plasma concentration (Cmax), area under the curve (AUC), half-life (t1/2) and assessment of translational biomarkers in plasma, PBMC's and tumor biopsies. Gene expression profiling of tumor tissue.
Time Frame: Cycle 1 and Cycle 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Arm 1: Carboplatin/Paclitaxel + Birinapant | Arm 2: Irinotecan + Birinapant | Arm 3: Docetaxel + Birinapant | Arm 4: Gemcitabine + Birinapant | Arm 5: Liposomal Doxorubicin + Birinapant
Serious Adverse Events (participants affected / at risk) | 9/24 | 41/83 | 16/33 | 13/18 | 9/18
Other Adverse Events (participants affected / at risk) | 24/24 | 83/83 | 33/33 | 18/18 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Carboplatin/Paclitaxel + Birinapant (N=24) | Arm 2: Irinotecan + Birinapant (N=83) | Arm 3: Docetaxel + Birinapant (N=33) | Arm 4: Gemcitabine + Birinapant (N=18) | Arm 5: Liposomal Doxorubicin + Birinapant (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 2 | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 5 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 3 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 5 | 0 | 2 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 4 | 5 | 1 | 1
Generalized oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 3 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cholangitis suppurative (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 5 | 2 | 1
Sepsis (Infections and infestations) | 1 | 4 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 5 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 8 | 1 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 4 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 | 1 | 2
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0
Caecitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 5 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Carboplatin/Paclitaxel + Birinapant (N=24) | Arm 2: Irinotecan + Birinapant (N=83) | Arm 3: Docetaxel + Birinapant (N=33) | Arm 4: Gemcitabine + Birinapant (N=18) | Arm 5: Liposomal Doxorubicin + Birinapant (N=18)
Anaemia (Blood and lymphatic system disorders) | 16 | 35 | 13 | 11 | 4
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 8 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 23 | 10 | 7 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 28 | 7 | 8 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 5 | 6 | 4 | 3 | 2
Ventricular extrasystoles (Cardiac disorders) | 2 | 2 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Arcus lipoides (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 1 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 3 | 1 | 4 | 0 | 0
Vision blurred (Eye disorders) | 1 | 2 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 4 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 32 | 5 | 5 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 9 | 5 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 7 | 4 | 2 | 3
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 10 | 25 | 15 | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 58 | 12 | 5 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 7 | 4 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 6 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 3 | 1 | 1
Flatulence (Gastrointestinal disorders) | 0 | 5 | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 1 | 2 | 2
Gingival pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 14 | 62 | 16 | 9 | 11
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 4 | 3 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 11 | 5 | 4 | 2
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 47 | 9 | 10 | 7
Asthenia (General disorders) | 9 | 23 | 10 | 7 | 5
Catheter site reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 3 | 0 | 0 | 1
Chills (General disorders) | 6 | 14 | 4 | 2 | 2
Device occlusion (General disorders) | 1 | 5 | 2 | 1 | 0
Disease progression (General disorders) | 0 | 4 | 5 | 1 | 1
Early satiety (General disorders) | 0 | 3 | 2 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 17 | 57 | 21 | 13 | 13
Generalized oedema (General disorders) | 0 | 2 | 1 | 1 | 0
Influenza like illness (General disorders) | 1 | 1 | 1 | 1 | 0
Infusion related reaction (General disorders) | 3 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 2 | 10 | 2 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 1
Oedema peripheral (General disorders) | 9 | 28 | 15 | 9 | 9
Pain (General disorders) | 2 | 3 | 2 | 1 | 0
Pyrexia (General disorders) | 6 | 16 | 6 | 8 | 4
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 3 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 6 | 5 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 2 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 3 | 1 | 2
Rhinitis (Infections and infestations) | 2 | 6 | 3 | 1 | 0
Sepsis (Infections and infestations) | 1 | 4 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 3 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 12 | 3 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 5 | 1 | 3 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 3 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 4 | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 6 | 2 | 2 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 6 | 1 | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 8 | 0 | 3 | 2
Blood creatinine increased (Investigations) | 3 | 11 | 3 | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 7 | 5 | 2 | 3
Blood urea increased (Investigations) | 3 | 5 | 3 | 2 | 1
Blood uric acid increased (Investigations) | 0 | 3 | 2 | 1 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 2 | 0 | 0
Breath sounds abnormal (Investigations) | 2 | 4 | 6 | 2 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 8 | 4 | 2 | 1
Haptoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Heart rate irregular (Investigations) | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 7 | 2 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 6 | 1 | 1 | 0
Occult blood positive (Investigations) | 1 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 4 | 4 | 0 | 2 | 0
Pulmonary percussion test abnormality (Investigations) | 0 | 0 | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 1 | 0
Urine bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 0 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Urine output increased (Investigations) | 0 | 0 | 0 | 0 | 1
Urobilinogen urine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 2 | 1 | 0
Weight decreased (Investigations) | 4 | 16 | 3 | 4 | 3
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 1
White blood cell count decreased (Investigations) | 2 | 10 | 0 | 1 | 0
White blood cell count increased (Investigations) | 3 | 3 | 2 | 1 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 10 | 42 | 15 | 8 | 7
Dehydration (Metabolism and nutrition disorders) | 4 | 31 | 6 | 3 | 5
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 6 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 6 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 9 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 7 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 20 | 8 | 7 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 6 | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 12 | 6 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 5 | 3 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 10 | 7 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 11 | 5 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 3 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 5 | 6 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 4 | 3 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 2 | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 11 | 17 | 2 | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 6 | 6 | 1 | 1
Extensor plantar response (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 14 | 1 | 5 | 3
Hyporeflexia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 3 | 1 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 3 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 7 | 1 | 7 | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 3 | 9 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2 | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Restless leg syndrome (Nervous system disorders) | 2 | 1 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Tardive dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 5 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 7 | 2 | 3 | 0
Confusional state (Psychiatric disorders) | 1 | 7 | 3 | 1 | 1
Depression (Psychiatric disorders) | 4 | 2 | 6 | 2 | 0
Hallucination (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 10 | 1 | 0 | 3
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 2 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 4 | 0 | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 2 | 0 | 2 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 3 | 2 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 4 | 3 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 19 | 7 | 5 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 4 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 3 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 5 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 5 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 1 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 34 | 8 | 0 | 3
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 7 | 2 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 4 | 2 | 2 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 9 | 3 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 16 | 4 | 4 | 2
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 5 | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 2 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 4 | 1 | 1 | 3
Flushing (Vascular disorders) | 4 | 2 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 5 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Hypotension (Vascular disorders) | 3 | 12 | 6 | 2 | 4
Orthostatic hypotension (Vascular disorders) | 2 | 2 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No